CLINICAL TRIAL: NCT01126957
Title: Combined Ketamine/Propofol for Emergency Department Procedural Sedation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left institution.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Project Number: 1084480
Record Dates: First submitted 2010-05-11; First posted 2010-05-20 (Estimated); Results first posted 2017-05-30 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-03

CONDITIONS: Procedural Sedation and Analgesia
MeSH Terms: conditions — Agnosia | interventions — Ketamine; Fentanyl; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Participants received 0.5-1.5 micrograms/kg Fentanyl, followed 0.5 mg/kg Ketamine infusion, followed by propofol to maintain sedation.
  Interventions: Drug: Ketamine; Drug: Fentanyl; Drug: Propofol
- Placebo (Placebo Comparator): Participants received 0.5-1.5 micrograms/kg Fentanyl, followed by placebo infusion, followed by propofol to maintain sedation.
  Interventions: Drug: Placebo; Drug: Fentanyl; Drug: Propofol

INTERVENTIONS:
Drug: Ketamine — Ketamine was given as a 0.5mg / Kg bolus.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Placebo — Placebo given as an bolus to control group.
  Arms: Placebo
Drug: Fentanyl — Fentanyl 0.5 - 1.5 micrograms given to both arms prior to Ketamine or placebo
  Other Names: Sublimaze
Drug: Propofol — Propofol given to both arms to maintain sedation throughout procedure.
  Other Names: Diprivan

SUMMARY:
Introduction

Numerous drugs and combinations of drugs are used for procedural sedation and analgesia (PSA) in Emergency Departments, including propofol, ketamine, benzodiazepines, narcotics, barbiturates, and others, but propofol has gained popularity despite its potential to cause cardiac and respiratory depression. Obviously the optimal agent or combination of agents has not been identified. There are reasons to believe that a combination of ketamine and propofol may have advantages over other agents/combinations. These include better hemodynamic stability at equal depth of anesthesia with a combination of ketamine/propofol than with propofol alone, less respiratory depression with the combination in comparison to propofol alone, and preservation of respiratory drive with the combination. There is one study of ketamine/propofol in Emergency Department (ED) procedural sedation which demonstrated the safety and effectiveness of the combination, but did not compare it to any other agents or combinations. The investigators designed a randomized, placebo controlled study to compare propofol to propofol and ketamine for adequacy of sedation and respiratory depression in Emergency Department procedural sedation and analgesia. The investigators hypothesis was that the combination of propofol/ketamine would produce better sedation and/or less respiratory depression than propofol alone.

Methods

Study design

The investigators conducted a randomized, prospective, double-blinded study of all patients receiving procedural sedation. From April 2007 until July 2009 in the ED of a 274 bed university teaching hospital. The study was approved by the University of Missouri's Institutional Review Board and informed consent was obtained from all participants.

DETAILED DESCRIPTION:
Introduction

Numerous drugs and combinations of drugs are used for procedural sedation and analgesia (PSA) in Emergency Departments, including propofol, ketamine, benzodiazepines, narcotics, barbiturates, and others, but propofol has gained popularity despite its potential to cause cardiac and respiratory depression. Obviously the optimal agent or combination of agents has not been identified. There are reasons to believe that a combination of ketamine and propofol may have advantages over other agents/combinations. These include better hemodynamic stability at equal depth of anesthesia with a combination of ketamine/propofol than with propofol alone, less respiratory depression with the combination in comparison to propofol alone, and preservation of respiratory drive with the combination. There is one study of ketamine/propofol in Emergency Department (ED) procedural sedation which demonstrated the safety and effectiveness of the combination, but did not compare it to any other agents or combinations. We designed a randomized, placebo controlled study to compare propofol to propofol and ketamine for adequacy of sedation and respiratory depression in Emergency Department procedural sedation and analgesia. Our hypothesis was that the combination of propofol/ketamine would produce better sedation and/or less respiratory depression than propofol alone.

Methods

Study design

We conducted a randomized, prospective, double-blinded study of all patients receiving procedural sedation. From May 2007 until March 2009 in the ED of a 274 bed university teaching hospital. The study was approved by the University of Missouri's Institutional Review Board and informed consent was obtained from all participants.

Study setting and population

All patients requiring PSA in the ED were viewed as potential subjects unless they were pregnant, less than 1 year of age, history of prior adverse reaction to anesthesia, underlying cardiac or pulmonary disease, hepatic dysfunction, porphyria, psychiatric illness, allergy to eggs/soybeans, increased intracranial or intraocular pressure, abnormal airway pathology or an American Society of Anesthesiologists (ASA) score of 3 or greater. The attending ED physician would then approach the patient to enroll them in the study. If the patient accepted they were randomized by the hospital pharmacy.

Study protocol

An ED attending physician was dedicated to PSA throughout the procedure. Patients had EKG, blood pressure, respiratory rate, pulse oximetry, and end-tidal carbon dioxide (PetCO2) monitored, had IV access obtained and were placed on nasal cannula oxygen supplementation. All patients received pre-procedure analgesia with 0.5 to 1.5 mcg/Kg of fentanyl and all patients had reflective sunglasses placed so as to obscure eye movements from the staff.

Subjects were randomized by the pharmacy in blocks of ten. Consecutively numbered pre-filled 3cc syringes were prepared by the pharmacy staff once they received a signed and dated study enrollment sheet from the ER staff with the patients weight in kilograms provided. All physicians, nurses, patients and study personnel were blinded to the contents of the syringes which were hand delivered by pharmacy personnel.

Patients were randomized to receive either 0.5 mg/Kg of ketamine or placebo (normal saline) delivered to the emergency room sedating physician in a 3 cc syringe containing a clear/colorless solution. This solution was delivered intravenously over a one minute infusion. On completion of this infusion all patients received propofol starting at 1 mg/Kg over 2 minutes and supplemented with repeated boluses of 0.5 mg/Kg to maintain adequate sedation. Patients were felt to be adequately sedated once they received a Colorado Behavioral Numerical Pain Scale (CBNPS) score of 0 to 113(table 1.) Patients were monitored after the procedure until a normal level of consciousness was observed.

The quantity of all drugs delivered were recorded. During the procedure all patients were monitored for 5 respiratory depression markers:

* PetCO2 rise of ³ 5 mm/Hg
* Respiratory rate < 8 br/min
* arterial oxygen saturation (SaO2) < 90%
* Apnea ³ 15 seconds
* Airway manipulation

Physicians were permitted to intervene and provide any supportive/resuscitative measures at there discretion despite the pre-specified respiratory depression markers.

All data were collected and recorded on standardized Hospital PSA forms. Data was collected for the entire time frame of the individual procedural sedations. Following the completion of the procedural sedation a second form was filled out by both the sedating physician and monitoring nurse recording specifically any respiratory events/rescue interventions and overall satisfaction with the procedural sedation. The overall quality of the PSA was evaluated by the physician/nurse performing the sedation as one of the following:

1. Not satisfied
2. Somewhat satisfied
3. Satisfied
4. Very satisfied
5. Excellent

All data was recorded on a secure computer in spreadsheet form (Microsoft Excel 2003, Microsoft Corporation, Redmond, WA) for later analysis.

Outcome Measures

Four endpoints were defined prior to study initiation:

Respiratory Depression. A difference in evidence of respiratory depression between the groups. Respiratory depression was defined as the occurrence of any of the 5 markers.

Satisfaction with PSA. A difference in the evaluation of the quality of the sedation by the providers.

Quality of PSA. Number of patients with a CBNPS of 0.

Propofol usage. Did the addition of ketamine significantly reduce the amount of propofol needed to produce adequate PSA.

Data analysis We plan to enroll 100 patients in each group. This is based on an estimate of a 40% incidence of respiratory depression with propofol alone, a reduction to 20% with the combination of ketamine/propofol, an a of 0.05 and a power of 0.8.14-16. An interim analysis was conducted at enrollment of 100 patients using a significance of 0.025 for difference in respiratory depression.

Respiratory depression and CBNPS were compared using a chi-squared test and Satisfaction with PSA and Quality of PSA were compared using a t-test. Tests were done with Primer of Biostatistics (Version 6.0, Stanton A. Glantz, 2005).

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals from 1 year of age and up without the below exclusion criteria

Exclusion Criteria:

* Subjects: All patients who require ED conscious sedation and do not meet any of the following exclusion criteria are eligible for study participation:

  * Age < 1yr
  * History of prior adverse reaction to anesthesia
  * History of cardiac disease
  * History of pulmonary disease
  * Hepatic dysfunction
  * Thyroid disease
  * Pregnancy
  * Porphyria
  * Psychiatric Illness
  * Allergy to eggs, soybeans, or sulfites
  * Increased intracranial or intraocular pressure
  * Active upper respiratory infection in children
  * Abnormal airway
  * ASA score of III or greater

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2007-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry David, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri - Columbia dept. of Emergency Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 107 participants were consented for the study. 103 completed.
Pre-assignment Details: We know that 107 participants had enrolled as of February 2008 and that 4 were terminated by the PI as not eligible. 103 were noted to have completed. However, the PI left the institution without making available any results or analyzed data.
Groups:
- Ketamine or Placebo: Participants received 0.5-1.5 micrograms/kg Fentanyl, followed 0.5 mg/kg Ketamine or placebo infusion, followed by propofol to maintain sedation.
  Ketamine: Ketamine was given as a 0.5mg / Kg bolus.
  Fentanyl: Fentanyl 0.5 - 1.5 micrograms given to both arms prior to Ketamine or placebo
  Propofol: Propofol given to both arms to maintain sedation throughout procedure.
Period: Overall Study
Arm/Group | Ketamine or Placebo
Started | 103
Completed | 103
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 107 participants signed the consent but 4 were found ineligible. 103 participants started and completed the study. Data were collected but not analyzed as the investigator left the institution prior to analysis and did not make data available for others to analyze.
Groups:
- Ketamine or Placebo: Participants received 0.5-1.5 micrograms/kg Fentanyl, followed 0.5 mg/kg Ketamine infusion or placebo, followed by propofol to maintain sedation.
  Ketamine: Ketamine was given as a 0.5mg / Kg bolus.
  Fentanyl: Fentanyl 0.5 - 1.5 micrograms given to both arms prior to Ketamine or placebo
  Propofol: Propofol given to both arms to maintain sedation throughout procedure.
Arm/Group | Ketamine or Placebo
Number analyzed (Participants) | 107
Age, Customized [Count of Participants; unit: Participants]
  Age >1 year | 107
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male and Female | 107

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Depression
Description: 1. Endotracheal carbon dioxide (ETCO2) rise > 5mm/hg
  2. Arterial oxygen saturation (SaO2) <90%
  3. Respiratory rate (RR) < 8 br/min
  4. Apnea > 15 sec
  5. airway manipulation
Time Frame: Baseline and throughout procedure
Population: 103 participants completed the study. Data were collected but were not analyzed prior to the investigator leaving the institution, and neither did he make the data available for analysis.
Arm/Group | Ketamine or Placebo
Number analyzed (Participants) | 0

2. Secondary Outcome: Satisfaction With Procedural Sedation
Description: Score of 1 to 5 with 5 being completely satisfied and 1 being not satisfied at all was recorded by both the monitoring nurse and the physician performing the procedural sedation
Time Frame: 20 minutes
Population: as for outcome 1
Groups:
- Ketamine: Participants received 0.5-1.5 micrograms/kg Fentanyl, followed 0.5 mg/kg Ketamine infusion or placebo, followed by propofol to maintain sedation.
  Ketamine: Ketamine was given as a 0.5mg / Kg bolus.
  Fentanyl: Fentanyl 0.5 - 1.5 micrograms given to both arms prior to Ketamine or placebo
  Propofol: Propofol given to both arms to maintain sedation throughout procedure.
Arm/Group | Ketamine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For the duration of the procedure for which each participant required sedation.
Description: Adverse event data were not made available by the investigator prior to him leaving the institution.
Groups:
- Ketamine or Placebo: Participants received 0.5-1.5 micrograms/kg Fentanyl, followed 0.5 mg/kg Ketamine infusion or palcebo, followed by propofol to maintain sedation.
  Ketamine: Ketamine was given as a 0.5mg / Kg bolus.
  Fentanyl: Fentanyl 0.5 - 1.5 micrograms given to both arms prior to Ketamine or placebo
  Propofol: Propofol given to both arms to maintain sedation throughout procedure.
Arm/Group | Ketamine or Placebo
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
107 participants were consented for the study. 4 were terminated by the investigator as they received surgery and were no longer eligible.

No data were analyzed/available as the target number of 200 was not reached; the PI has left the institution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes